CLINICAL TRIAL: NCT05756179
Title: Clinical Study Evaluating the Effect of Diosmin and Hesperidin in Treatment of Patients With Rheumatoid Arthritis
Brief Title: Effect of Diosmin and Hesperidin in Treatment of Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201734
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Diosmin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Diosmin 450 mg and Hesperidin 50 mg Combination /tablet/ twice daily for 3 months + Conventional Therapy (Methotrexate)
  Interventions: Drug: Diosmin and Hesperidin Combination
- Control group (No Intervention): Conventional Therapy (Methotrexate) only

INTERVENTIONS:
Drug: Diosmin and Hesperidin Combination — Diosmin 450 mg and Hesperidin 50 mg Combination
  Other Names: Diosmin Plus 500 mg tablet
  Arms: Intervention group

SUMMARY:
Evaluating the effect of the flavonoids combination (diosmin and hesperidin) as adjuvant therapy on patients with rheumatoid arthritis

DETAILED DESCRIPTION:
Evaluation of the anti inflammatory and antioxidant effects of the flavonoids combination (diosmin and hesperidin) as adjuvant therapy on patients with rheumatoid arthritis.

Clinical and functional assessment of disease activity.

Evaluation of hepatoprotective effect against methotrexate induced liver adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate disease activity.
* Patient age must be more than 18 years.

Exclusion Criteria:

* Pregnant and lactating females.
* Patients with liver, renal impairment or any other inflammatory diseases.
* Patients on TNF-α (tumor necrosis factor- α) or IL-1β (interleukin-1β) antagonists.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Anti inflammatory Effect | 3 months
  Measure the change in serum level of IL-1β (interleukin 1β) at baseline and after treatment in both groups
Effect on disease activity | 3 months
  Measure the change in the disease activity at baseline and after 3 months of therapy for each patient in both groups using Disease Activity Score-CRP (DAS28-CRP) which is calculated by a computer based formula consists of several variables: number of swollen joints (0-28), number of tender joints (0-28) and C reactive protein (CRP) (mg/l).
  A DAS28 value of >5.1 indicates high disease activity, DAS28 ranged from 3.3 to 5.1 indicates moderate disease activity and DAS28 ≤3.2 indicates low disease activity.

SECONDARY OUTCOMES:
Hepatoprotective Effect | 3 months
  Measure the change in serum level of Liver enzymes (ALT & AST) at baseline and after treatment in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ABDELBAR, MSc, Principal Investigator — College of Pharmacy - Arab Academy for Science and Technology; AHMED ELMALLAH, PhD, Study Chair — Faculty of Pharmacy - Alexandria University; MANAL TAYEL, MD, Study Chair — Faculty of Medicine - Alexandria Univeristy; ABEER IBRAHIM, MD, Study Chair — Faculty of Medicine - Alexandria Univeristy; NOHA HAMDI, PhD, Study Director — Faculty of Pharmacy - Alexandria University
Locations (1):
- Alexandria university hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No